CLINICAL TRIAL: NCT05462782
Title: Task Paired Transcranial Magnetic Stimulation for Working Memory Potentiation
Brief Title: TMS for Investigating Memory Facilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of sufficient personnel to run this study's research visits.
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00216935
Record Dates: First submitted 2022-06-17; First posted 2022-07-18 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Age-associated Memory Impairment
Keywords: Transcranial Magnetic Stimulation; Paired Associative Stimulation; Working Memory; Older adults; Functional Magnetic resonance imaging
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to understand how Transcranial Magnetic Stimulation(TMS) synchronized with a memory event can enhance working memory capacity. For this purpose, we will synchronize hippocampal directed stimulation, primary motor cortex stimulation and sham stimulation at Inter Stimulus Interval (ISI) 200 and 0 ms. The effects on memory will be assessed by a working memory task and resting state functional MRI .
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): Older healthy participants will be scanned with MRI and undergo memory task synchronized PAS with an active TMS in each visit with different stimulation localization and ISIs.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) Cone Coil
- Sham TMS (Sham Comparator): Older healthy participants will be scanned with MRI and undergo memory task synchronized PAS with a sham TMS coil in each visit with different ISIs application.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) Sham Coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) Cone Coil — The cone coil Cool-DB80 (MagPro, MagVenture, Alpharetta GA, US) will be used with an MRI-based TMS navigation system (Localite, St Augustin, Germany). TMS interventions will involve the following parameters: 1. Hippocampal directed stimulation at ISI 0ms, 2. Hippocampal directed stimulation at ISI 200ms, 3. Motor cortex stimulation at ISI 0ms, and 4. Motor cortex stimulation at ISI 200ms.
  Arms: Active TMS
Device: Transcranial Magnetic Stimulation (TMS) Sham Coil — The sham coil Cool B65 A/P (MagPro, MagVenture, Alpharetta GA, US) will be used with an MRI-based TMS navigation system (Localite, St Augustin, Germany). The different TMS interventions will be involve the following parameters: 1. Sham stimulation at ISI 0ms, and 2. Sham stimulation at ISI 200ms.
  Arms: Sham TMS

SUMMARY:
The aim of this study is to investigate the effects of Transcranial Magnetic Stimulation (TMS) following a Paired Associative Stimulation (PAS) protocol on the memorization capacity of elderly individuals. For this purpose, we will apply TMS synchronized with a working memory (WM) task and assess its effects on cortical connectivity and memorization capacity by Magnetic Resonance Imaging (MRI) and WM task learning. This study will be carried out in an older population of healthy participants. We will use the study results to refine the task related PAS protocol towards enhancing memory performance and brain connectivity.

DETAILED DESCRIPTION:
The fundamental objective is to evaluate the changes derived from the specific Paired Associative Stimulation (PAS) protocol applying Transcranial Magnetic Stimulation (TMS) towards the hippocampus to enhance memory in an older population. We will evaluate the following effects: 1) Changes in memory capacity using task performance of the working memory (WM) task and calculating the correctly memorized items; and 2) Changes in brain connectivity using resting state functional Magnetic Resonance Imaging (rs-fMRI) and comparing the correlated activity between areas related to the process of memorization.

In order to understand the memory and brain connectivity changes derived from the PAS intervention more specifically, we will characterize the stimulation localization, the Inter Stimulus Interval (ISI) timing and rule out training and placebo effects. To research if the PAS effects are specific to the stimulated brain area, we will conduct a control group in which stimulation will be delivered to the primary motor area (M1). Then, we will compare the outcome measures (changes in memory capacity and brain connectivity) between the different brain areas. To characterize the ISI, our goal is to calculate the synchronization timing that triggers cortical plastic changes. Thus, we will test two different ISI between the TMS pulse delivery and memorization task. Finally, to differentiate the effects that are derived from the PAS versus the effects from repetition of the task or placebo effects, we will conduct another control group with Sham TMS stimulation and reproduce the same experimental procedures as the group that receives the TMS stimulation. Sham TMS is used in this study to compare if brain stimulation (active TMS) can help improve memory compared to receiving no brain stimulation (sham TMS).

ELIGIBILITY:
Inclusion Criteria for Older Healthy Participants:

* Age from 60 to 85 years, inclusive (For piloting purposes, this inclusion criteria may vary).
* No history of a brain and/or skull lesion (e.g., stroke)
* Normal vision (can be corrected)
* Able to understand and give informed consent
* No neurological disorders
* Able to understand and speak English

Exclusion Criteria for Healthy Participants:

* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
* Surgical clips in the head or previous neurosurgery
* Any magnetic particles in the body
* Cochlear implants
* Prosthetic heart valves
* Epilepsy or any other type of seizure history
* History of significant head trauma (i.e., extended loss of consciousness, neurological sequelae)
* Significant claustrophobia
* Ménière's disease
* Pregnancy or breast feeding
* Non prescribed drug use
* History of current substance abuse (exception: current nicotine use is allowed)
* Marijuana
* Any neurological diagnoses
* Dementia; severe depression; or prior neurosurgical procedures
* Tremor or parkinsonism, or psychiatric disease that would interfere with study procedures for TMS, or MRI.
* Significant other disease (cardiological or heart disease, renal, hepatic, malignant tumors, mental or psychiatric disorders) that would prevent participants from fully engaging in study procedures
* Prisoners
* Medications contraindicated for TMS: antipsychotic and antidepressant medications.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Changes in Working Memory (WM) capacity | Compared during each visit between baseline, immediately after the intervention, and 30 minutes after intervention
  The WM task utilized is a customized version of the masking task model, presented by Sana Inoue and Tetsuro Matsuzawa, in 2007. This task is organized in three phases: 1) Waiting phase: a visual cue is presented to indicate the initiation of the trial; 2) Coding and retention phase: numbers are presented in a random arrangement within a 5x5 square matrix; and 3) Recall phase: the numbers disappear, leaving a white background as a clue, and the subject completes the task by pressing the squares in the matrix following the incremental order of the numbers. (Figure 2). The task ends either when the subject makes a mistake or completes correctly selecting all numbers in incremental order. The outcome measure for WM capacity is the amount of correctly remembered items (hit items) of each trial.
Changes in resting state functional MRI connectivity | Compared during each visit between baseline and 30 minutes after intervention
  The neural connectivity index that we will assess responds to the strength of synaptic connections between neurons and over time. The identification of correlations between remote brain areas will be tested by resting state functional magnetic resonance imaging (rs-fMRI). We will compare the connectivity network after intervention time with baseline and sham group. Correlations of spontaneous modulations in the blood oxygen level dependent (BOLD) signal will be analyzed and regions with similar functional properties under resting conditions will be detected. This analysis is able to identify significant long-lasting effects of active stimulation (vs. sham) on brain connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, Ph.D, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Only authorized personal listed on this IRB will have access to the data. During and after the study, all study records will be assigned a unique subject identifier code to protect the confidentiality of the participant's personal information. The information will be labeled with an unidentifiable code to reduce the risks to participant privacy. Once research information has been collected, we may share some of it. Any research information shared with people outside of Shirley Ryan AbilityLab/Northwestern University will not contain the participant's name, address, telephone or social security number, or any other direct personal identifier unless disclosure of the direct identifier is required by law.